CLINICAL TRIAL: NCT06446401
Title: Longitudinal Evaluation of Adding Docetaxel to ADT and Novel Hormone Treatment for Patients With High Volume Metastatic Hormone Sensitive Prostate Cancer in Order to Assess Relative Effectiveness: the Case of "Triple" Versus "Double" Therapy
Brief Title: The Case of "Triple" Versus "Double" Therapy for Patients With High Volume Metastatic Hormone Sensitive Prostate Cancer
Acronym: Lead4Care
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); University Hospital, Umeå (Other); Sahlgrenska University Hospital (Other); Saint Göran Hospital (Unknown); Swedish Cancer Society (Other); Uddevalla Hospital (Unknown); Östersund Hospital (Unknown); Ryhov County Hospital (Other); Mälarsjukhuset Hospital, Eskilstuna (Unknown); Västmanlands Hospital, Västerås, Sweden (Unknown); Gävle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01881-02
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; mHSPC; Comparative effectiveness evaluation; Triple therapy; Double therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Triple therapy: Patients with mHSPC and high tumour burden receiving treatment with androgen deprivation treatment, new hormone therapy (abiraterone, apalutamide, enzalutamide or darolutamide) and docetaxel.
  Interventions: Drug: ADT + NHT + Docetaxel
- Double therapy: Patients with mHSPC and high tumour burden receiving treatment with androgen deprivation treatment and new hormone therapy (abiraterone, apalutamide, enzalutamide or darolutamide).
  Interventions: Drug: ADT + NHT

INTERVENTIONS:
Drug: ADT + NHT + Docetaxel — Lead4Care leaves the treatment choice to the clinicians and the patients, i.e., does not intervene in their choice of treatment. However, Lead4Care proxy a randomized controlled experiment in which the intervention would be to add docetaxel to androgen deprivation treatment, new hormone therapy (abiraterone, apalutamide, enzalutamide or darolutamide). This involves a comparison of triple and double therapies. This group recives the triple therapy, i.e. ADT, NHT and Docetaxel.
  Groups: Triple therapy
Drug: ADT + NHT — Lead4Care leaves the treatment choice to the clinicians and the patients, i.e., does not intervene in their choice of treatment. However, Lead4Care proxy a randomized controlled experiment in which the intervention would be to add docetaxel to androgen deprivation treatment, new hormone therapy (abiraterone, apalutamide, enzalutamide or darolutamide). This involves a comparison of triple and double therapies. This group recives double therapy, i.e. they are receiving NHT and ADT, but not Docetaxel.
  Groups: Double therapy

SUMMARY:
Lead4Care is an observational, open-label, multicenter study evaluating the effectiveness, tolerance, and cost-effectiveness of triple against double therapy in matched groups of mHSPC patients with high tumor burden. In addition to androgen deprivation therapy (ADT), the triple constitutes of docetaxel and novel hormonal therapy (NHT), and the double of NHT therapy in addition to ADT.

Their effectiveness is compared in terms of mortality and morbidity, which is captured by HRQoL, pain, fatigue. Potential side effects are captured by neuropathy, diarrhea, constipation, anxiety, sickness, and dyssomnia. The cost-effectiveness is evaluated within a Markov model from a societal perspective in which the main disease stages are mHSPC, mCRPC and death.

In connection with a regular visit in hospital care, prostate cancer patients who in addition to ADT will initiate double or triple therapy are offered participation in the study. If the patient consent on-line, the patient will receive 13 online surveys over a 60-month period. The surveys are sent with an interval of two months for the first six months, quarterly thereafter until two years, and thereafter yearly.

Once all participants have been recruited, the baseline data shared by healthcare personnel and patients will be enriched with registry data. This baseline and registry data involves information about the patients' historical and current health- and socioeconomic status. Thereby, Lead4Care will be able to identify comparable groups of patients on triple and double treatments by using advanced matching methods.

In order to assure an objective analysis, Lead4Care will not allow any data extraction until Lead4Care has predefined and published all details regarding the comparison. The existing protocol is then complemented with a more detailed description of the comparison groups, the hierarchy of outcomes, and the analysis methods for these outcomes.

For these treatments, the main objectives are to:

* Compare mortality and morbidity on triple and double therapy, and their relative side-effects.
* Capture patient preferences for these different treatment outcomes over time.
* Evaluate cost-effectiveness of triple versus double therapy from a societal perspective.

DETAILED DESCRIPTION:
Comprehensive evaluation:

The treatment landscape of metastatic hormone-sensitive prostate cancer (mHSPC) is evolving rapidly and treatment guidelines often need to be made before the effectiveness of available combinations have been compared. Such is the case for the current recommendation to combine androgen deprivation therapy (ADT) with new hormonal therapy (NHT) and docetaxel (DTX). This triple therapy has not yet been directly evaluated against the alternative of ADT and NHT, i.e., the double therapy. The therapies have only been evaluated indirectly in the trials PEACE-1 and ARASENS. Lead4Care will evaluate triple against double therapy with regard to potential differences in disease progression as well as tolerance. Thereby, Lead4Care will do a comprehensive comparative effectiveness (CE) evaluation which can contribute to the pool of evidence important for future guidelines.

Observational design:

Lead4Care leaves the treatment choice to the clinicians and the patients, and uses advanced matching methods to ensure comparability between patients receiving triple- and double therapy. As the groups are expected to differ in terms of their tolerance to DTX, and the doctors valuation of tolerance differ, Lead4Care expect to be able to identify such matching groups on a subset of enrolled patients. The matched groups will be used for the CE evaluation. Patients will consequently be enrolled and followed prospectively irrespective of which therapy the clinicians will choose, and similar groups will be matched especially with regard to their tolerance to DTX as proxied by their age, comorbidity, ECOG collected within Lead4Care but also in terms of their health- and socioeconomic status (SES) in general requested from national registries. The matched groups will be as similar as expected in a randomized experiment in terms of tolerance in particular, but also in terms of health, and SES. Consequently, there is no need for randomization to ensure comparability, using this study design.

Lean observational design:

The additional data that prospective studies usually collect from healthcare, can pose an administrative burden on healthcare workers. Lead4Care has therefore invested considerable effort in developing the study design which leaves few tasks to healthcare workers, i.e., only screen the patient population and report the baseline data. Instead, Lead4Care will take responsibility for all future contact with the patients according to the study protocol. This involves supporting patients in consenting to the study and in reporting their symptoms, tolerance, and progressions in the 13 on-line questionnaires. The patients will hold a patient paper diary with such critical information that the study ask the patients to remember from healthcare visits, i.e., the date and levels for PSA:s, the date for castration resistant, and the date for next treatment. Lead4Care will therefore test a design that minimizes the burden on healthcare systems and which could remove some of the administrative barriers for CE evaluations.

Pain focus:

Recent research suggests that improved pain awareness could potentially reduce the risk of SREs and/or mortality. The rationale behind this is that pain seems to serve as an indicator of development of bone metastasis as the disease advances. Adequate disease management and properly pain control can help mitigate skeleton-related events (SRE), which, in turn, can impact mortality rates. For that reason, Lead4Care will evaluate pain differences across the treatments, and explore how these pain differences potentially can predict SRE and/or mortality.

Cost-effective care:

In Sweden, the cost for prostate cancer consumes a considerable part (12%) of our cancer related healthcare costs, which in in turn constitute 3% of the total healthcare costs. Choosing cost-effective prostate cancer treatments could consequently have a visible impact on Swedish healthcare costs. Lead4Care will therefore evaluate the triple- against the double therapy from a health-economic perspective. The additional cost for adding DTX and treating its potential complications (neurotoxicity, GI side-effects, osteoporosis etc.) will be compared against the difference in quality adjusted life years (QALY). This ratio is used within Sweden for prioritization of scarce resources. Lead4Care can therefore serve as a model for the health-economic (HE) evaluations, which becomes increasingly important as the availability of prostate cancer treatments is increasing.

Patient-centered care:

In healthcare, there is often a dilemma since treatments for prostate cancer can provide survival benefits for the patients but at potential HRQoL loss. For instance, patients who undergo surgery improve their survival but their HRQoL may worsen because of complications. Moreover, patients who receive DTX in the triple therapy may improve their survival but their HRQoL may worsen because of side-effects. Lead4Care has therefore developed an instrument together with patients which captures patients treatment preferences. This instrument will ascertain patients' preferences for life prolonging or HRQoL improving treatments. Lead4Care will therefore help us better understand the populations treatment preferences. This information is important in order to better take the patients preferences into account in planning their care, just as is required in the Swedish Patient Act.

Objectives:

With the implementation of Lead4Care, the hope is to achieve the following objectives:

To evaluate the clinical effectiveness of triple- versus double therapy in matched groups of mHSPC patients with high tumour burden.

To evaluate the tolerance of triple- versus double therapy in matched groups of mHSPC patients with high tumour burden.

To describe the patients treatment preferences (gain in survival against loss of HRQoL) for mHSPC patients with high tumour burden.

To describe the cost-effectiveness of adding DTX for mHSPC-patients with high tumour burden.

To evaluate the clinical effectiveness of triple- versus double therapy in matched sub-groups of mHSPC patients with high tumour burden (e,g, w/wo visceral metastases).

To explore the way pain proxy for or predict SRE and survival for mHSPC-patients with high tumour burden with baseline bone metastases.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all of the following criteria:

* Patients should have initiated triple or double therapy no longer than 3 months from the start of ADT,
* Patients must have mHSPC at the time of enrolment, and high metastatic burden.
* Patients must be ≥ 18 years old at the time of enrolment. Note: NHT could be abiraterone acetate, apalutamide, darolutamide or enzalutamide.

Exclusion Criteria:

Participants meeting any of the of the following criteria are not eligible for inclusion:

* Patients who do not understand written and/or oral instructions in Swedish.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mHSPC and high tumor burden initiating treatment with triple or double therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | : Measured at month 2, 4, 6, 9, 12, 15, 18, 21, 24, 36, 48, 60 and thereafter annually until month 144 (12 years).
  Death due to any causes, i.e., overall survival (OS). captured by the Swedish National Cause of Death Register.

SECONDARY OUTCOMES:
Fatigue | Measured at baseline and month 2, 4, 6, 12, 18, 24, 36, 48 and 60.
  Fatigue is a PROM captured by FACIT-F fatigue domain, PGI-C and 3 additional questions related to different aspects of fatigue added by the researchers.
  FACIT-F fatigue domain contains 13 questions regarding fatigue. The respondent is asked to report how much the respondent agrees with different statements, measured on a scale between Not at all (0) and Very much (4).
  Patient Global Impression of Fatigue Change (PGI-C) is included to understand if the fatigue differences across the treatments are clinically significant. Thereby, the Minimal Important Differences (MIDs) for the different fatigue measurements can be derived. PGI-C is reported on a 7-grade scale, ranging from Very large deterioration (0) to Very large improvement (6).
  Other questions:
  VAS-scale ranging between No fatigue (0) and Worst possible fatigue (100) Present fatigue, ranging from No fatigue (0) to Excruciating (5). Worst fatigue last 3 weeks, ranging from No fatigue (0) to Excruciating (5)
Time to progression | Measured at month 2, 4, 6, 9, 12, 15, 18, 21, 24, 36, 48 and 60.
  Time until the patients' prostate cancer becomes castration resistant (mCRPC) is based on patient-reported survey data regarding their progression.
Time to first line treatment of mCRPC | Measured at month 2, 4, 6, 9, 12, 15, 18, 21, 24, 36, 48, 60 and thereafter annually until month 144 (12 years).
  Time until the patient receives first line treatment for mCRPC is captured by patient reported survey data regarding their start of first line treatment for their mCRPC stage.
Pain intensity | Measured at baseline and month 6, 12, 18, 24, 36, 48, and 60.
  Pain is a PROM captured by The McGill Pain Questionnaire and 3 additional questions related to different aspects of pain added by the researchers.
  McGill contains 15 questions regarding type of pain, reported on a 4-grade scale between None (0) and Severe (3). It also contains a VAS-scale ranging between No pain (0) and Worst possible pain (100), as well as a question of present pain intensity, ranging from No pain (0) to Excruciating (5).
  Patient Global Impression of Pain Change (PGI-C) has been included to understand if the pain differences across the treatments are clinically significant. Thereby, the Minimal Important Differences (MIDs) for the different pain measurements can be derived. PGI-C is reported on a 7-grade scale, ranging from very large deterioration (0) to very large improvment.
  Other questions Yes/No question if the participants experience any pain. 2 questions regarding placement and type of pain.

OTHER OUTCOMES:
Skeleton Related Events (SRE) | Measured at month 2, 4, 6, 9, 12, 15, 18, 21, 24, 36, 48, 60 and thereafter annually until month 144 (12 years).
  SRE measured through Swedish registers and is assumed to have occurred if the patient experiences a hospitalization due to a pathologic fracture (ICD codes M485, M495, M844 and M907) or spinal cord compression (ICD codes G550, G834, G952, G958, G959 and G992).
General Health-Related Quality of life (HRQoL) | Measured at baseline and month 2, 4, 6, 9, 12, 15, 18, 21, 24, 36, 48 and 60.
  HRQoL is a patient reported outcome measurement captured by EuroQol's 5Q-5D-5L and 1 additional question added by the researchers.
  EQ-5D-5L contains 5 questions regarding the patients HRQoL measured on a 5-grade scale where lower scores indicates better health. It also includes a VAS-scale ranging between Worse possible health (0) and Best possible health (100).
  The researchers have added a question regarding the overall health of the participant, measured on a 5-grade scale where lower scores indicates better health.
Side effects | Measured at baseline and month 2, 4, 6, 9, 12, 15, 18, 21, 24 36, 48 and 60.
  Side effects is a patient reported outcome measurement captured by FACT-GOG-NTX domain and 7 additional questions developed by the researchers relating to GI-symptoms, sleep disturbances, nervous tensions (anxiety) and medical infections. The additional questions are measured on a 5-grade scale, ranging from No day (1) to Every day (5).
  FACT-GOG-NTX domain contains 11 questions related to neuropathy and how much the respondent agrees with different statements, measured on a scale between Not at all (0) and Very much (4).
Prostate cancer specific health-related quality of life (PC-HRQoL) | Measured at baseline and month 6, 12, 18, 24, 36, 48 and 60.
  PC-HRQoL is a PROM captured by FACT-P and PGI-C.
  FACT-P contains 5 domains and 39 questions regarding different aspects of HRQoL. The respondent is asked to report how much they agree with different statements on a scale between Not at all (0) and Very much (3).
  Patient Global Impression of HRQoL Change (PGI-C) is included to understand if the HRQoL differences across the treatments are clinically significant. Thereby, the Minimal Important Differences (MIDs) for the different HRQoL measurements can be derived. PGI-C is reported on a 7-grade scale, ranging from Very large deterioration (0) to Very large improvement (6).
Treatment preferences trade-off | Measured at baseline and month 6, 12, 18, 24, 36, 48 and 60.
  This instrument measures the patient tolerance for HRQoL deterioration in order to increase life expectency.
  The respondent is first asked to state his current HRQoL in a VAS-scale ranging between No HRQoL (0) and Full HRQoL (100). The respondent is then asked if he has any absolute preferences for either HRQoL or length of life. If the respondent has no such absolute preference, he is asked to state how much HRQoL deterioration he would tolerate for an increased life expectency of 6 months.
  The instrument has been developed in collaboration with patients along with input from researchers and healthcare professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Langenskiöld, SRLECT & PhD, Principal Investigator — Uppsala University
Locations (2):
- Sweden (2):
  - Uppsala University Hospital, Uppsala, Region Uppsala
  - Uppsala University, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: Undecided